CLINICAL TRIAL: NCT04892355
Title: Postoperative Pain After İntracanal Procedures Based On Different İrrigation Activation Tecniques: A Randomized, Clinical Trial
Brief Title: Postoperative Pain After İntracanal Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Yahya Güven, Assist. Prof. Dr. Yahya GÜVEN, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AfyonkarahisarHSU
Record Dates: First submitted 2021-05-11; First posted 2021-05-19 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Endodontically Treated Teeth
Keywords: EDDY; EndoActivatör; Xp-endo Finisher; Postoperative pain
MeSH Terms: conditions — Tooth, Nonvital; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: 4-group clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Conventional Syringe Irrigation Group (Experimental): During the final irrigation procedure, a 30 - G side vented needle was placed 2 mm shorter than the working length and was applied without agitation. 5 mL of 2.5% NaOCl was applied for 1 minute for each channel. Each canal was then washed with 2 mL of 17% EDTA for 1 minute.
  Interventions: Device: Root canal irrigation
- Xp Endo Finisher Group (Experimental): Xp Endo Finisher file was used with VDW Silver (VDW) endomotor at 800 rpm speed and 1 Ncm torque according to the manufacturer's instructions. The Xp Endo Finisher file was placed in the canal, 2 mm shorter than the working length, and was used with slow movements of 7-8 mm amplitude in the canal during activation. 5 mL of 2.5% NaOCl was applied for 1 minute for each channel. Each canal was then washed with 2 mL of 17% EDTA for 1 minute.
  Interventions: Device: Root canal irrigation
- EDDY Group (Experimental): An EDDY tip of size 25/04 was used for sonic activation. The EDDY was placed in the duct 2 mm shorter than the working length and the activation process was performed with slow movements with an amplitude of 2-4 mm. In the irrigation process, 5 mL of 2.5% NaOCI was applied for 1 minute for each channel. Each canal was then washed with 2 mL of 17% EDTA for 1 minute.
  Interventions: Device: Root canal irrigation
- Endoactivator Group (Experimental): Medium Endoactivator tip of 25 / .04 size was used for irrigation activation. Medium type was placed in the canal 2 mm shorter than the working length and activation was performed by making short strokes of 2-3 mm. 5 mL of 2.5% NaOCl was applied for 1 minute for each channel. Each canal was then washed with 2 mL of 17% EDTA for 1 minute.
  Interventions: Device: Root canal irrigation

INTERVENTIONS:
Device: Root canal irrigation — Devices used during root canal irrigation
  Other Names: EndoActivator (Dentsply Tulsa Dental Specialties, Tulsa, OK)-XP-endo Finisher (XPF; FKG Dentaire SA, La Chaux-de-Fonds, Switzerland)- EDDY (EDDY; VDW, Munich, Germany)-

SUMMARY:
Aim: The aim of this study is to investigate the effects of different irrigation activation systems on pain after endodontic treatment in molar teeth with irreversible pulpitis.Post-operative pain values of the participants will be recorded and evaluated with the VAS scale.

Postoperative pain values of the techniques will be compared with statistical evaluation.

DETAILED DESCRIPTION:
Aim: The aim of this study is to investigate the effects of different irrigation activation systems on pain after endodontic treatment in molar teeth with irreversible pulpitis.Materials and Methods: The study will be carried out on 140 patients with molar teeth diagnosed with irreversible pulpitis. After the root canal preparation is completed, the patients will be divided into 4 groups according to the irrigation activation system; Conventional syringe irrigation (CSI), EDDY, EndoActivator (EA) and Xp-endo Finisher (XPF). After the irrigation process is completed, the root canals will be filled using gutta-percha and canal sealer and the treatment will be completed in one session. Pain values at 6, 24, 48, 72 hours and 7 days after treatment will be evaluated at a 0.05% significance level using the Kruskal-Wallis test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients ranging between 18 and 60 years in age
* Patients that experienced moderate-to-severe pain represented on a visual analogue scale (VAS)
* Maxillar and Mandibular molar teeth were diagnosed with symptomatic irreversible pulpitis

Exclusion Criteria:

* Any systemic disease and pregnancy in the patient
* Having used analgesic-anti-inflammatory in the last 12 hours and cortisone for the last 6 months
* The patient has bruxism
* Teeth with severe damage
* Teeth with calcified canals
* Teeth with pain to percussion
* Teeth with periapical radiolucency
* Teeth with root resorption
* Teeth with an immature / open apex
* Teeth with previous RCT

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — No gender discrimination will be applied in the study.
Enrollment: 140 (Estimated)
Dates: Start 2022-08-06 (Estimated); Primary Completion 2022-10-06 (Estimated); Study Completion 2022-11-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain After İntracanal Procedures Based On Different İrrigation Activation Tecniques: A Randomized, Clinical Trial | one week(7 days)
  Preoperative pain of the patients before the treatment was recorded with the VAS scale. Pain levels were classified as 0: no pain, 1-3: mild pain, 4-6: moderate pain, 7-10: severe pain .After the treatment of the patients, a pain assessment form was given to the patient in order to evaluate the postoperative pain. Patients were asked to mark their pain levels on the VAS scale. The marking procedure was taught to the patients by a blinded researcher from the groups. When the patients came to the control appointment, VAS scales were collected and the data were analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: yahya güven, Principal Investigator — Afyonkarahisar Health Sciences University